CLINICAL TRIAL: NCT03385850
Title: The Roles of Th17/Treg Cells and IL-23/IL-17 Axis in the Mechanisms of Early Enteral Nutrition Improving Immune Function of Sepsis
Brief Title: The Th17/Treg Cells and IL-23/IL-17 Axis and Early Enteral Nutrition in Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, XiangWang, Director, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NanjingFirst
Record Dates: First submitted 2017-12-14; First posted 2017-12-29 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Sepsis; Immune System Disorder; Enteral Feeding
MeSH Terms: conditions — Sepsis; Immune System Diseases | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early enteral nutrition (Experimental)
  Interventions: Other: enteral nutrition
- delayed enteral nutrition (Active Comparator)
  Interventions: Other: enteral nutrition

INTERVENTIONS:
Other: enteral nutrition — early enteral nutrition group or delayed enteral nutrition group

SUMMARY:
The investigators aim to evaluate the roles of Th17/Treg cells and IL-23/IL-17 axis in the mechanisms of early enteral nutrition (EEN) correcting immune imbalance of sepsis by means of improving the intestinal flora disturbance. The results of this study would lay the foundation for revealing the mechanisms of EEN improving immune imbalance of sepsis and provide a new idea to the early treatment of sepsis

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of sepsis
2. Within 3 days of sepsis onset before ICU admission
3. No artificial nutrition (enteral or parenteral nutrition) were provided before ICU admission

Exclusion Criteria:

1. Ileus
2. Digestive tract hemorrhage
3. Inflammatory bowel disease
4. Abdominal hypertension (IAP >25mmHg)
5. Cancer or chronic organ dysfunction (e.g., hepatic or renal dysfunction)
6. Malnutrition or immunodeficiency
7. Long-term use of hormones

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
28-d mortality | 28 days

SECONDARY OUTCOMES:
immune parameters | 7 days
  serum Th17 and Treg lymphocyte percentages
immune parameters | 7 days
  IL-23, IL-17, IL-6, IL-10 levels

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
There is a plan to make individual participant data (IPD) available to other researchers.